CLINICAL TRIAL: NCT01278875
Title: High Density Lipoprotein Function in Acute Coronary Syndromes
Brief Title: Function of High Density Lipoproteins in Acute Coronary Syndromes
Acronym: HDL_ACS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Jacques Genest, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 10-208-BMA
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Acute Coronary Syndrome
Keywords: High density lipoproteins; Acute coronary syndromes; Cellular cholesterol efflux; HDL: proteomics; Nitric Acid production
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Plasma HDL isolated by ultracentrifugation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acute Coronary Syndrome: Subjects with ACS within 72 hours of clinical presentation
- Stable CAD subjects: Patients with stable, chronic CAD
- Control subjects: Healthy individuals

SUMMARY:
High density lipoproteins (HDL) have many effects that protect against cardiovascular diseases. In an acute heart attack (acute coronary syndrome -ACS), HDL change in composition and structure, reflecting the inflammatory environment that accompanies an ACS. The investigators will examine the function of HDL during an ACS and again when the patient has recovered.

DETAILED DESCRIPTION:
High density lipoproteins (HDL) have pleiotropic effects associated with protection against atherosclerosis. These effects include cellular cholesterol efflux, anti-inflammatory and anti-oxidant effects, increase in nitric acid (NO) production from vascular endothelial cells and differentiation of endothelial progenitor cells for repair at sites of vascular injury. The measurement of the cholesterol mass within HDL (HDL-C) does not provide an adequate measure of HDL function. The investigators therefore propose to test and validate biomarkers of HDL function in patients with acute coronary syndromes (ACS).

Hypothesis: HDL lose their cardiovascular protective functions in ACS. The investigators hypothesize that these changes are transient and partly normalize within 12 weeks. In this proposal, the investigators will examine the function of HDL in acute coronary syndromes (ACS) and 12 weeks later, in the recovery phase. Acute coronary syndromes are characterized by an acute inflammatory reaction, a marked decrease in HDL in plasma and a shift of the HDL proteome to an inflammatory phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-80 years of age
* Acute Coronary Syndrome within 72 hours of presentation
* Elevated tropinins (T or I)

Exclusion Criteria:

* Refusal to participate
* Inability to return for a 12 week follow-up visit
* Hemodynamic instability requiring vasopressor support, mechanical ventricular assist devices, the need for coronary artery bypass surgery
* Lack of documented atherosclerotic CAD
* Uncontrolled hypertension
* Triglycerides≥5mmol/L
* Severe obesity (BMI≥35)
* Alcohol intake>21 drinks/week
* Presence of thyroid, hepatic, or renal disease
* Autoimmune disease or any chronic or acute infectious or inflammatory illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to hospital with an acute coronary syndrome, within 72 hours
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2011-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
HDL-mediated cellular cholesterol efflux | 12 weeks
  Biomarkers of HDL function

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Genest, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada